CLINICAL TRIAL: NCT00388063
Title: A Phase II Open-Label Study of the Safety and Efficacy of Atiprimod Treatment for Patients With Low to Intermediate Grade Neuroendocrine Carcinoma
Brief Title: Safety and Efficacy of Atiprimod Treatment for Patients With Low to Intermediate Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Callisto Pharmaceuticals (Industry)
Responsible Party: Gary Jacob, Callisto Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-106; WIRB 20061681
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Neuroendocrine Carcinoma
Keywords: Neuroendocrine; Carcinoma; Atiprimod; Carcinoid
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoma; Carcinoid Tumor | interventions — azaspirane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atiprimod — oral, 14 days on / 14 days off; 30mg capsules

SUMMARY:
This study will evaluate the safety and efficacy of atiprimod treatment in patients with low to intermediate grade neuroendocrine carcinoma who have metastatic or unresectable local-regional cancer and who have either symptoms (diarrhea, flushing and/or wheezing) despite standard therapy (octreotide) or progression of neuroendocrine tumor(s).

DETAILED DESCRIPTION:
For carcinoid, despite the many cytotoxic chemotherapy trials that have been conducted, no regimen has demonstrated a response rate of more than 20% using the criterion of a 50% reduction of bidimensionally measurable disease. In the more recently reported ECOG phase III study of chemotherapy in carcinoid tumors (E1281), patients were randomly assigned to treatment with 5-fluorouracil (5FU) plus doxorubicin or 5FU plus streptozocin. The median progression free survival durations were disappointing. They were 4.5 months in the 5FU plus doxorubicin arm and 5.3 months in the 5FU plus streptozocin arm. Overall survival durations recorded in the trial were also suboptimal at 15 and 24 months respectively. There is no clear survival benefit for cytotoxic chemotherapy.

This is a phase II, multi-center, open-label study of the safety and efficacy of atiprimod treatment in patients with low to intermediate grade neuroendocrine carcinoma who have metastatic or unresectable local-regional cancer and who have either symptoms (diarrhea, flushing and/or wheezing) despite standard therapy (octreotide) or progression of neuroendocrine tumor(s) (defined as the appearance of one or more new lesions or a 20% increase in the sum of the longest diameter of target lesions during the 6 months prior to enrollment). A maximum of 40 evaluable patients will be enrolled in this study. Atiprimod will be administered orally as a single daily dose of 120 mg/day for 14 days, followed by a 14-day treatment-free period (i.e., 1 treatment cycle = 28 days).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have documented histologic proof of low or intermediate grade neuroendocrine carcinoma. Both carcinoid (any site; atypical/intermediate grade carcinoid is allowed) and islet cell (pancreatic endocrine tumor) will be eligible. Patient with neuroendocrine tumors associated with MEN1 syndrome will be eligible.
* Patients must have either metastatic or unresectable local-regional cancer. Patients with brain metastases are allowed on study, but they must have evaluable target lesions elsewhere.
* Patients must have measurable disease, as defined by RECIST.
* Patients must have either symptoms (diarrhea, flushing and/or wheezing) despite standard therapy (octreotide) or progression of neuroendocrine tumor(s) (defined as the appearance of one or more new lesions or a 20% increase in the sum of the longest diameter of target lesions during the 6 months prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction of symptoms (diarrhea, flushing and/or wheezing) | 1 year
Progression of neuroendocrine tumor(s) | 1 year

SECONDARY OUTCOMES:
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary Jacob, Ph.D., Study Director — Callisto Pharmaceuticals
Locations (8):
- United States (8):
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Cedars Sinai Outpatient Cancer Center at the Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Scott and White Memorial Hospital, Scott Sherwood and Brindley Facility, Temple, Texas